CLINICAL TRIAL: NCT00271661
Title: Presbyopia in Breast Cancer Survivors
Status: Withdrawn | Type: Observational
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Other Study IDs: BR-1-0072; ETHICS 22007
Record Dates: First submitted 2005-12-30; First posted 2006-01-04 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Presbyopia
Keywords: presbyopia; breast cancer survivors
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Chemotherapy drugs, used in cancer treatments, may change the timing of a vision condition known as presbyopia. Presbyopia is the inability to focus the eye on close objects, by a process called accommodation. It is caused by an increase in the stiffness of the lens of the eye that occurs naturally with aging. Currently, there are no known treatments that can be used to prevent or delay presbyopia. As a result, the risk, in later life, of having this condition is essentially 100%.

The purpose of this research is to determine whether chemotherapy drugs are delaying the age at which people develop symptoms of presbyopia. We hope to establish that presbyopia can in fact be delayed with the use of drugs, which would ultimately lead to further research in this area.

DETAILED DESCRIPTION:
Chemotherapy drugs, used in cancer treatments, may change the timing of a vision condition known as presbyopia. Presbyopia is the inability to focus the eye on close objects, by a process called accommodation. It is caused by an increase in the stiffness of the lens of the eye that occurs naturally with aging. Currently, there are no known treatments that can be used to prevent or delay presbyopia. As a result, the risk, in later life, of having this condition is essentially 100%.

The purpose of this research is to determine whether chemotherapy drugs are delaying the age at which people develop symptoms of presbyopia. We hope to establish that presbyopia can in fact be delayed with the use of drugs, which would ultimately lead to further research in this area.

ELIGIBILITY:
Inclusion Criteria:

* ages 45-60
* ability to understand and provide written consent in English

Exclusion Criteria:

* blindness
* visual defects leading to accommodative failure
* severe myopia
* recurrent breast cancer

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-08; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Overall Officials: John Mackey, Dr., Principal Investigator — AHS Cancer Control Alberta